CLINICAL TRIAL: NCT02716454
Title: Early Surgery Versus Conservative Treatment in Patients With Ileocaecal Crohn's Disease - Prospective Randomized Study
Brief Title: Early Surgery Versus Conservative Treatment in Patients With Ileocaecal Crohn's Disease
Acronym: ESPRIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ondrej Ryska (Other)
Responsible Party: Sponsor-Investigator, Ondrej Ryska, investigator secretary in section of IBD surgery Czech Surgical Society, Czech Surgical Society
Organization: Czech Surgical Society (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBDchirCZ-01
Record Dates: First submitted 2016-03-17; First posted 2016-03-23 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Crohn's Disease
Keywords: Early surgery; Crohn's disease; Step-up therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Surgery - ES (Experimental): Early laparoscopic ileocaecal resection
  Interventions: Procedure: Ileocaecal resection
- Step-up therapy - STUP (No Intervention): Treatment with step-up conservative approach according to good clinical practice.

INTERVENTIONS:
Procedure: Ileocaecal resection — laparoscopic ileocaecal resection with primary anastomosis
  Arms: Early Surgery - ES

SUMMARY:
This study compares the efficacy of early surgical with medical treatment in patients with ileocaecal uncomplicated Crohn's disease. The patients with affected short part of terminal ileum will be randomized either for laparoscopic ileocaecal resection or standard step-up pharmacological therapy.

DETAILED DESCRIPTION:
Surgical therapy is currently indicated for Crohn's disease (CD) patients after conservative treatment becomes ineffective. The principles of so-called step-up therapy (STUP) where surgery represents the last therapeutical option are still followed.

Early surgical intervention (Early Surgery - ES) can be an alternative even in patients with uncomplicated type of CD before all medical therapy is used (Top-down approach). Limited resection under these conditions will lead to immediate remission. Moreover, laparoscopic ileocaecal resection is safe with low morbidity and regarding potential complications of step-up treatment might be beneficial for the patient.

Before wide introduction of ES approach into clinical practice, it is necessary to perform a randomized trial comparing early resection with the standard step-up medical therapy.

The potential effect of early, intensive therapy (ileocaecal resection) on biological behavior of the disease has not been studied that is why patients with uncomplicated ileocaecal form are the most suitable for such a trial. Significant number of these patients will indeed progress into more unfavorable course of the disease (relapse, complicated form, early recurrence).

Other potential benefit of early resection is the extended period without necessary medication. Even pharmacological recurrence prevention is not needed after surgery in uncomplicated CD patient if other risk factors are excluded. Rapid remission induced by surgery can lead to faster improvement of quality of life than long-term medication.

ELIGIBILITY:
Inclusion criteria

* All patients aged 18-65 years with a uncomplicated ileocaecal form of Crohn's disease (affected < 20 cm of terminal ileum) (type: L1B1) diagnosed within last 12 months
* Diagnose confirmed by endoscopy including appropriate extent of disease and presence of ulcers in terminal ileum
* Patient is able to understand the study and sign an informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Previous bowel resection or other extensive abdominal surgery, which primarily excludes laparoscopic approach
* Affected other parts of the digestive tract or symptomatic stenosis or stenosis impassable for the endoscope or presence of prestenotic dilatation in terminal ileum confirmed by enterography
* Any extraluminal complications of Crohn's disease (fistula, abscess)
* Affected part of terminal ileum longer than 20 cm
* Severe comorbidities (heart failure, renal failure, liver failure, severe disorders of the central and peripheral nervous system, serious infectious disease) or patient with ASA (American Society of Anesthesiologists) III and more
* Malnutrition or presence of another serious risk factor, which contradicts construction of primary anastomosis
* Current use of immunosuppressive or biologic therapy

Other exclusion criteria:

* Different intraoperative finding
* Protocol violation
* Subject refuses further participation in the study
* Termination of the trial by responsible authority

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2021-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Endoscopic remission | 24 months
  The rate of endoscopic remission defined as Rutgeerts score ≤ 1 and SES-CD = 0 in early surgery and standard step-up therapy group respectively

SECONDARY OUTCOMES:
QoL | 24 months
  Quality of life measured by IBDQ, IBD Disability index
Clinical remission | 24 months
  Clinical remission defined by Crohn's disease activity index < 150
Drug consumption | 24 months
  Overall drug consumption (corticosteroids, antibiotics, immunomodulators, biologic therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Ondrej Ryska, Dr, PhD, Principal Investigator — Section of IBD surgery - Czech Surgical Society
Locations (12):
- Czechia (12):
  - The University Hospital Brno, Brno
  - Hospital Ceske Budejovice, České Budějovice
  - Horovice Hospital, Hořovice
  - Universitiy Hospital Hradec Kralove, Hradec Králové
  - Hospital Jihlava, Jihlava
  - Hospital Liberec, Liberec
  - Vitkovice Hospital, Ostrava - Vitkovice
  - University Hospital in Pilsen, Pilsen
  - Royal Vinohrady University Hospital, Prague
  - Institute for Clinical and Experimental Medicine, Prague
  - Na Homolce Hospital, Prague
  - ISCARE, Prague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jess T, Riis L, Vind I, Winther KV, Borg S, Binder V, Langholz E, Thomsen OO, Munkholm P. Changes in clinical characteristics, course, and prognosis of inflammatory bowel disease during the last 5 decades: a population-based study from Copenhagen, Denmark. Inflamm Bowel Dis. 2007 Apr;13(4):481-9. doi: 10.1002/ibd.20036. PMID 17206705
- [Background] Domenech E, Zabana Y, Garcia-Planella E, Lopez San Roman A, Nos P, Ginard D, Gordillo J, Martinez-Silva F, Beltran B, Manosa M, Cabre E, Gassull MA. Clinical outcome of newly diagnosed Crohn's disease: a comparative, retrospective study before and after infliximab availability. Aliment Pharmacol Ther. 2010 Jan 15;31(2):233-9. doi: 10.1111/j.1365-2036.2009.04170.x. Epub 2009 Oct 13. PMID 19832727
- [Background] Cosnes J, Nion-Larmurier I, Beaugerie L, Afchain P, Tiret E, Gendre JP. Impact of the increasing use of immunosuppressants in Crohn's disease on the need for intestinal surgery. Gut. 2005 Feb;54(2):237-41. doi: 10.1136/gut.2004.045294. PMID 15647188
- [Background] Golovics PA, Lakatos L, Nagy A, Pandur T, Szita I, Balogh M, Molnar C, Komaromi E, Lovasz BD, Mandel M, Veres G, Kiss LS, Vegh Z, Lakatos PL. Is early limited surgery associated with a more benign disease course in Crohn's disease? World J Gastroenterol. 2013 Nov 21;19(43):7701-10. doi: 10.3748/wjg.v19.i43.7701. PMID 24282358
- [Background] Eshuis EJ, Bemelman WA, van Bodegraven AA, Sprangers MA, Bossuyt PM, van Milligen de Wit AW, Crolla RM, Cahen DL, Oostenbrug LE, Sosef MN, Voorburg AM, Davids PH, van der Woude CJ, Lange J, Mallant RC, Boom MJ, Lieverse RJ, van der Zaag ES, Houben MH, Vecht J, Pierik RE, van Ditzhuijsen TJ, Prins HA, Marsman WA, Stockmann HB, Brink MA, Consten EC, van der Werf SD, Marinelli AW, Jansen JM, Gerhards MF, Bolwerk CJ, Stassen LP, Spanier BW, Bilgen EJ, van Berkel AM, Cense HA, van Heukelem HA, van de Laar A, Slot WB, Eijsbouts QA, van Ooteghem NA, van Wagensveld B, van den Brande JM, van Geloven AA, Bruin KF, Maring JK, Oldenburg B, van Hillegersberg R, de Jong DJ, Bleichrodt R, van der Peet DL, Dekkers PE, Goei TH, Stokkers PC. Laparoscopic ileocolic resection versus infliximab treatment of distal ileitis in Crohn's disease: a randomized multicenter trial (LIR!C-trial). BMC Surg. 2008 Aug 22;8:15. doi: 10.1186/1471-2482-8-15. PMID 18721465
- [Background] Rutgeerts P, Geboes K, Vantrappen G, Beyls J, Kerremans R, Hiele M. Predictability of the postoperative course of Crohn's disease. Gastroenterology. 1990 Oct;99(4):956-63. doi: 10.1016/0016-5085(90)90613-6. PMID 2394349
- [Background] Peyrin-Biroulet L, Cieza A, Sandborn WJ, Coenen M, Chowers Y, Hibi T, Kostanjsek N, Stucki G, Colombel JF; International Programme to Develop New Indexes for Crohn's Disease (IPNIC) group. Development of the first disability index for inflammatory bowel disease based on the international classification of functioning, disability and health. Gut. 2012 Feb;61(2):241-7. doi: 10.1136/gutjnl-2011-300049. Epub 2011 Jun 5. PMID 21646246
- [Background] Dignass A, Van Assche G, Lindsay JO, Lemann M, Soderholm J, Colombel JF, Danese S, D'Hoore A, Gassull M, Gomollon F, Hommes DW, Michetti P, O'Morain C, Oresland T, Windsor A, Stange EF, Travis SP; European Crohn's and Colitis Organisation (ECCO). The second European evidence-based Consensus on the diagnosis and management of Crohn's disease: Current management. J Crohns Colitis. 2010 Feb;4(1):28-62. doi: 10.1016/j.crohns.2009.12.002. Epub 2010 Jan 15. No abstract available. PMID 21122489
- [Background] Maartense S, Dunker MS, Slors JF, Cuesta MA, Pierik EG, Gouma DJ, Hommes DW, Sprangers MA, Bemelman WA. Laparoscopic-assisted versus open ileocolic resection for Crohn's disease: a randomized trial. Ann Surg. 2006 Feb;243(2):143-9; discussion 150-3. doi: 10.1097/01.sla.0000197318.37459.ec. PMID 16432345
- [Result] Aratari A, Papi C, Leandro G, Viscido A, Capurso L, Caprilli R. Early versus late surgery for ileo-caecal Crohn's disease. Aliment Pharmacol Ther. 2007 Nov 15;26(10):1303-12. doi: 10.1111/j.1365-2036.2007.03515.x. Epub 2007 Sep 10. PMID 17848181